CLINICAL TRIAL: NCT06209190
Title: Safety and Feasibility of Total Marrow and Total Lymphoid Irradiation as Conditioning Regimen in Allogeneic Hematopoietic Stem-cell Transplantation
Brief Title: Safety and Feasibility of TMLI as Conditioning Regimen in Allogeneic Hematopoietic Stem-cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Head of hematology, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Safety TMLI in HSCT
Record Dates: First submitted 2023-08-31; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Our study will enroll 14 patients in an estimated period of 2 years, with non-probabilistic sampling based on consecutive cases from January 2022 to January 2024 based on prior local transplant data. The study will be done according with the Declaration of Helsinki, and with Good Clinical Practice guidelines and the protocol will be approved by local Institutional Review Board after external review and will be locally funded.
  Descriptive statistics will be used to report the baseline variables of the patients. Groups will be compared with hypothesis tests through deductive statistics using Student's t test or Mann Whitney U test accordingly, to determine significant differences between two groups and their means; and the Chi square test as a verification test and comparison of hypotheses of categorical data, in addition, survival analysis will be carried out by the Kaplan-Meier method and competing risk analysis as appropriate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total marrow and lymphoid irradiation (TMLI) (Experimental): TMLI will be added in doses of 12 Gy on days -3 to -1 divided into 6 fractions of 2 Gy every 12 hours for 3 days, which will be administered through a computed tomography tomotherapy system.
  Interventions: Radiation: total marrow and total lymphoid irradiation

INTERVENTIONS:
Radiation: total marrow and total lymphoid irradiation — doses of 12 Gy on days -3 to -1 divided into 6 fractions of 2 Gy every 12 hours for 3 days, which will be administered through a computed tomography tomotherapy system plus conditioning scheme of our institution

SUMMARY:
Multiple conditioning regimens have been used for the HSCT, some of which include radiotherapy. Total body irradiation (TBI) has demonstrated to be superior to chemotherapy alone in the phase III FORUM trial. However, concerns for long-term toxicity have made TBI less used. Total marrow and lymphoid irradiation (TMLI) has emerged as a new alternative that can potentially keep the benefits of radiation but reducing toxicity to healthy tissues.

The primary objective of this trial is to evaluate the feasibility and safety of TMLI as part of conditioning schemes with or without etoposide for HSCT in patients between age 16 and 45 years with ALL in first line or relapsed disease. As secondary endpoint the efficacy will be assessed by minimal residual disease at 60 days post-transplant, as well as other outcome measures such as non-relapse mortality (NRM), relapse free survival (RFS) and overall survival (OS).

DETAILED DESCRIPTION:
TMLI will be administered as part of the conventional reduced intensity conditioning scheme of our institution:

Fludarabine 25 mg/m2 + cyclophosphamide 350 mg/m2 on days -6 to -3, for patients with positive measurable residual disease TMLI will be added in doses of 12 Gy on days -3 to -1 divided into 6 fractions of 2 Gy every 12 hours for 3 days, which will be administered through a computed tomography tomotherapy system.

Infusion of peripheral blood hematopoietic stem cells will be performed on day 0 and after this, prophylaxis for GVHD with post-transplant cyclophosphamide 50 mg/kg will be administered on days +3 and +4, followed by tacrolimus or cyclosporine A plus mycophenolate mofetil regardless of HLA matching.

The procedure for the donation of hematopoietic cells will be done through a peripheral blood apheresis with previous stimulation with filgrastim at 10 mcg/kg for 4 days according to the standardized procedures of our institution.

The leukocyte and platelet count will be monitored by serial complete blood count, and a bone marrow aspiration (BMA) and minimal residual disease (MRD) will be performed on day 60 after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALL confirmed by flow cytometry.
* Patients between age 16 and 45 years with ALL in first remission, refractory, or relapsing
* Patients who have an identical or haploidentical allogeneic donor by high resolution HLA

Exclusion Criteria:

* Patients who do not meet the age previously mentioned.
* Patient with comorbidities that rule them out for HSCT, with a Hematopoietic cell transplantation-specific comorbidity index (HCT-CI) greater than 2.
* Poor performance status or Karnofsky less than 70%
* Transthoracic echocardiogram with alteration in myocardial function with left ventricular ejection fraction (LVEF) less than 50%
* Patients who previously and for another reason have already received radiotherapy or who refuse to receive it

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Early mortality rate | 30 days
  Primary outcome of safety will be determined by early mortality rate (before day +30) with an expected rate lower than 15%.
Serious adverse events | 30 days
  Co-primary outcome will be the appearance of serious adverse effects (grade equal to or higher than 3) according to the common terminology criteria for adverse events of the US National Cancer Institute (NCL-CTCAE v.5).

SECONDARY OUTCOMES:
Measurable residual disease | 60 days
  Measurable residual disease assessment through flow cytometry in bone marrow aspirate
Non-relapse mortality | 12 months
  Event of death in patients without disease relapse with death after relapse as a competing risk.
Event-free survival | 12 months
  Survival without event of disease progression, relapse or death after enrollment.
Overall survival | 12 months
  Survival time after enrollment
Graft versus host disease incidence | 12 months
  Incidence of graft versus host disease according to MAGIC and NIH criteria

CONTACTS AND LOCATIONS:
Overall Officials: David R Gomez-Almaguer, MD, Study Chair — Universidad Autonoma de Nuevo Leon
Locations (1):
- Andres Gomez, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stein A, Palmer J, Tsai NC, Al Malki MM, Aldoss I, Ali H, Aribi A, Farol L, Karanes C, Khaled S, Liu A, O'Donnell M, Parker P, Pawlowska A, Pullarkat V, Radany E, Rosenthal J, Sahebi F, Salhotra A, Sanchez JF, Schultheiss T, Spielberger R, Thomas SH, Snyder D, Nakamura R, Marcucci G, Forman SJ, Wong J. Phase I Trial of Total Marrow and Lymphoid Irradiation Transplantation Conditioning in Patients with Relapsed/Refractory Acute Leukemia. Biol Blood Marrow Transplant. 2017 Apr;23(4):618-624. doi: 10.1016/j.bbmt.2017.01.067. Epub 2017 Jan 10. PMID 28087456
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28087456/